CLINICAL TRIAL: NCT02488694
Title: A Randomized, Open-label, Phase II Study of Maintaining Pan-ERBB Blockade Following Platinum-based Induction Chemotherapy in Patients With EGFR Mutated, Metastatic Non-small-cell Lung Cancer Progressing After Treatment With Afatinib as First EGFR-targeting Agent
Brief Title: Maintaining ERBB Blockade in EGFR-mutated Lung Cancer
Acronym: MARBLE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unsufficient recruitment
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-TRK-0114
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Non-small-cell Lung Cancer With Somatic EGFR Mutations
MeSH Terms: interventions — Afatinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Afatinib (Experimental): 105 patients to be treated with afatinib
  Interventions: Drug: Afatinib
- Arm B: Pemetrexed (Active Comparator): 105 patients to be treated with pemetrexed
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Afatinib — 40 mg/d
  Other Names: GIOTRIF®
  Arms: Arm A: Afatinib
Drug: Pemetrexed — 500 mg/m² i.v. on d1 of each 21-day cycle
  Other Names: ALIMTA®
  Arms: Arm B: Pemetrexed

SUMMARY:
This study aims to compare the efficacy of afatinib maintenance with pemetrexed maintenance following induction therapy with platinum/ pemetrexed in patients with metastatic epidermal growth factor receptor (EGFR) mutated non-small-cell lung cancer (NSCLC) progressing after first-line treatment with afatinib with respect to progression-free survival.

DETAILED DESCRIPTION:
This is a randomized, open-label, phase II study of maintaining pan-ERBB blockade following platinum-based induction chemotherapy in patients with EGFR mutated, metastatic NSCLC progressing after first-line treatment with afatinib.

Patients who have progressed after first-line treatment with afatinib will be screened while receiving an induction phase which consists of at least three but not more than four cycles of cisplatin/carboplatin plus pemetrexed given in 21-day cycles. Patients who do not progress (i.e. complete or partial response, or stable disease - CR, PR or SD) after completion of three or four cycles induction chemotherapy will then be randomized (1:1 ratio) to receive maintenance therapy with either afatinib (40 mg/d, or last dose if reduced during first-line treatment) or pemetrexed (500 mg/m² every 21 days, or 375 mg/m² if dose was reduced during induction therapy) until disease progression, unacceptable toxicity or patient consent withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of non-small-cell lung cancer (NSCLC) with no curative therapeutic option. Patients with Stage IV (UICC 7th edition) disease or Stage IIIB disease not amenable to curative intent surgery or radiotherapy are enrolled. Patients with mixed histology are eligible if NSCLC is the predominant histology
2. Documented somatic EGFR mutation as determined by medically accepted assay technology
3. Patients with documented progression after response (CR/PR) or stable disease (SD) for at least 6 months of treatment with afatinib as first tyrosine kinase inhibitor (either given as first-line therapy or being switched to afatinib after up to 4 courses of platinum-based chemotherapy)
4. Patients who have completed 3 or 4 cycles of cisplatin or carboplatin plus pemetrexed induction chemotherapy prior to randomization leading to documented response (CR/PR) or SD according to RECIST 1.1
5. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
6. Male or female patient with age ≥18 years
7. ECOG performance status ≤ 2
8. Adequate organ and bone marrow function, defined as all of the following:

   Before the last cycle of induction chemotherapy or after hematopoietic recovery from the last cycle of induction chemotherapy:
   * Absolute neutrophil count (ANC) ≥ 1,500 / mm3
   * Platelet count ≥ 100,000 / mm3
   * Creatinine clearance ≥ 45 ml / min (calculated according to Cockroft and Gault, or Tc99m-DPTA clearance or similar methodology). Patients with creatinine clearance of 45 to 79 ml/min should refrain from using NSAID at least 2 days before and 2 days after infusion of pemetrexed. Long-acting NSAID should be terminated 5 days before pemetrexed infusion.
   * Total serum bilirubin ≤ 1.5 times upper limit of institutional normal (ULN)
   * Serum aspartate amino transferase (AST) and serum alanine amino transferase (ALT) ≤ 3 times the upper limit of institutional normal (ULN) ( ≤ 5 times ULN if liver function abnormalities are due to underlying malignancy)
9. Recovered from any previous therapy related toxicity to ≤ Grade 1 at study entry (except for stable sensory neuropathy ≤ Grade 2 and alopecia)
10. Written informed consent
11. Ability to comply with the protocol for the duration of the study, including hospital/office visits for treatment and scheduled follow-up visits and examinations

Exclusion Criteria:

1. Systemic therapy for metastatic disease or relapse other than (a) first-line therapy with afatinib or (b) afatinib given as first EGFR-targeting agent following up to 4 courses of platinum-based chemotherapy with no disease progression between first-line chemotherapy and initiation of afatinib (prior adjuvant chemotherapy is allowed) and 3 to 4 cycles of induction chemotherapy with cisplatin or carboplatin and pemetrexed following afatinib failure
2. Prior treatment with erlotinib, gefitinib or other investigational or approved EGFR-targeting small molecules or antibodies
3. Known EGFR T790M mutation (analysis not mandatory)
4. Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study
5. Extended radiotherapy within 4 weeks prior to randomization, except as follows:

   1. Palliative, limited local radiation to non-target lesions (e.g. isolated bone metastases) may be allowed up to 2 weeks prior to randomization, and
   2. single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling
6. Active brain metastases except for the followings:

   * Asymptomatic brain metastases incidentally found during screening process which do not require local treatment in the opinion of the investigator.
   * Asymptomatic brain metastases for which local treatment has been given: stable for at least 4 weeks of lower dose corticosteroids (e.g., dexamethasone up to 4 mg/d) and/or non-enzyme-inducing anti-convulsants treatment before study randomization.
   * Brain metastases controlled after surgery and/or radiotherapy
7. Meningeal carcinomatosis
8. Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, non-invasive bladder cancer, ductal carcinoma in situ of the breast, or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured. Definitively treated localized low/intermediate risk prostate cancer (Gleason score ≤ 7) is allowed when a rise in serum PSA level by ≥ 2 ng/mL above the nadir is excluded
9. Known pre-existing interstitial lung disease
10. Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug in the opinion of the investigator (e.g. Crohn's Disease, ulcerative colitis, chronic diarrhea, and malabsorption)
11. Clinically relevant cardiovascular abnormalities as judged by the investigator such as uncontrolled hypertension, congestive heart failure ≥ NYHA grade III, unstable angina or myocardial infarction within the past 6 months, or poorly controlled cardiac arrhythmia in the opinion of investigator
12. Any history of or concomitant condition that, in the opinion of the investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug, or renders the patient at high risk of treatment complications
13. Women of child-bearing potential and men who are able to father a child, unwilling to be abstinent or use adequate contraception prior to study entry, for the duration of study participation and for at least 2 weeks after treatment has ended
14. Female patient pregnant or breast-feeding
15. Known active infection with HBV, HCV or HIV
16. Any contraindications for therapy with pemetrexed
17. Known hypersensitivity to afatinib or the excipients of any of the trial drugs
18. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 60 days prior to treatment start
19. Pleurocentesis or paracentesis should be considered in patients with clinically significant pleural effusions or ascites if clinically indicated. However, per SmPC of pemetrexed the presence of effusion is not an exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 40 months
  The primary endpoint of this study is progression-free survival (RECIST 1.1).

SECONDARY OUTCOMES:
Overall survival | 40 months
  Efficacy measure
Objective response rate | 40 months
  Objective response rate (ORR), clinical benefit rate (RECIST 1.1); Efficacy measure
Quality of Life | 40 month
  Health-Related Quality of Life (HRQoL)
Safety (intensity and incidence of adverse events, graded according to US NCI CTCAE Version 4.03) | 40 month
  Safety, toxicity (intensity and incidence of adverse events, graded according to US NCI CTCAE Version 4.03)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schuler, Prof. Dr., Principal Investigator — Westdeutsches Tumorzentrum, Universitätsklinikum Essen
Locations (1):
- Universitätsklinikum Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Working Group for Medical Oncology (AIO) from the German Cancer Society (DKG) — http://www.aio-portal.de